CLINICAL TRIAL: NCT01888666
Title: Comparison Between Rapid and Slow Palatal Expansion: Evaluation of Periodontal Indices
Status: Completed | Type: Observational
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Enrico Marchetti, Contract professor, University of L'Aquila
Other Study IDs: Tecc01/2013
Record Dates: First submitted 2013-02-04; First posted 2013-06-28 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Palatal Expansion Technique

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- rapid palatal expansion (RPE) using the Haas appliance
- slow palatal expansion (SPE)

SUMMARY:
The aim of this study is to evaluate the periodontal effects during rapid palatal expansion (RPE) or slow palatal expansion (SPE) and to compare them by means of periodontal indices, in order to establish the possible differences and advantages of one of these treatments in periodontal terms.

Materials and methods: 10 patients will selected and submitted to RPE treatment; other 10 patients will selected and submitted to SPE treatment. The patients will treated with the Haas appliance. In both the groups the periodontal clinical indices (plaque index, PI; papillary bleeding index, PBI; probing pocket depth, PPD) will collected three times during the treatment (before, during and at the end). All measurements will performed by the same examiner.

A descriptive statistical analysis will conducted. The paired samples Student's T test will used to evaluate the intra-group differences between t1 and t2. The unpaired samples Student's T test will used to evaluate between groups differences at t1 and t2. The significance level will set at 95%.

ELIGIBILITY:
Inclusion Criteria:

* palate narrow
* necessity of performing a expansion treatment

Exclusion Criteria:

* dental disease

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients attending the division of orthodontics of Department MeSVA, University of L'Aquila, Italy
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
evaluation of periodontal health by probing pocket depth, PPD | Change from Baseline in probing pocket depth at 20 days and 5 months of active therapy
  In the Group I (RPE), probing pocket depth were detected in three stages:
  T0, detected 7 days after the periodontal prophylaxis (at the beginning of the active orthodontic therapy) ; T1, detected after 20 days of active therapy; T2, detected after 5 months of retention therapy.
  In the Group II, the collected data corresponded to:
  T0, detected 7 days after the periodontal prophylaxis; T1, detected during clinical control after 3 months of active therapy; T2, detected after 3 months of restraint. All measurements were performed by the same examiner.

SECONDARY OUTCOMES:
valuation of periodontal health by plaque index, PI | Change from Baseline in plaque index at 20 days and 5 months of active therapy
  In the Group I (RPE), plaque index were detected in three stages:
  T0, detected 7 days after the periodontal prophylaxis (at the beginning of the active orthodontic therapy) ; T1, detected after 20 days of active therapy; T2, detected after 5 months of retention therapy.
  In the Group II, the collected data corresponded to:
  T0, detected 7 days after the periodontal prophylaxis; T1, detected during clinical control after 3 months of active therapy; T2, detected after 3 months of restraint. All measurements were performed by the same examiner.
evaluation of periodontal health by papillary bleeding index, PBI | Change from Baseline in papillary bleeding index at 20 days and 5 months of active therapy
  In the Group I (RPE), papillary bleeding index were detected in three stages:
  T0, detected 7 days after the periodontal prophylaxis (at the beginning of the active orthodontic therapy) ; T1, detected after 20 days of active therapy; T2, detected after 5 months of retention therapy.
  In the Group II, the collected data corresponded to:
  T0, detected 7 days after the periodontal prophylaxis; T1, detected during clinical control after 3 months of active therapy; T2, detected after 3 months of restraint. All measurements were performed by the same examiner.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Life, Health and Environmental Science, University of L'Aquila, L’Aquila, AQ, Italy